CLINICAL TRIAL: NCT01649778
Title: PRINCIPAL: A Prospective Observational Study of Real World Treatment Patterns and Treatment Outcomes in Patients With Advanced or Metastatic Renal Cell Carcinoma Receiving Pazopanib
Brief Title: Observational Study of Real World Effectiveness Data and Safety in Patients Receiving Pazopanib With Advanced or Metastatic Renal Cell Carcinoma
Acronym: PRINCIPAL
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: 115232; CPZP034A2401 (Other: Novartis)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — Not applicable. This is a Non-interventional study collecting prospective observational data.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pazopanib: Prospective Observational study collecting real world data on Pazopanib in patients with advanced or metastatic Renal Cell Carcinoma. Study is considered non-interventional, no drug will be provided. No study visits or procedures are mandated per protocol.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Prospective Observational study collecting real world data on Pazopanib in patients with advanced or metastatic Renal Cell Carcinoma. Study is considered non-interventional, no drug will be provided. No study visits or procedures are mandated per protocol.
  Other Names: Votrient

SUMMARY:
This is a global, multi-centre, long-term, prospective, observational study to evaluate treatment patterns and clinical outcomes in patients with advanced or metastatic RCC treated for the first time with pazopanib. The study is designed to enroll approximately 700-1000 patients in over the course of an enrollment period of approximately 18 months.There are no protocol-mandated visits or procedures associated with the study. Each patient is expected to participate for a maximum of 30 months or until premature discontinuation (i.e., due to death, withdrawal of consent, lost to follow-up or study termination).

DETAILED DESCRIPTION:
This is a global, multi-centre, long-term, prospective, observational study to evaluate treatment patterns and clinical outcomes in patients with advanced or metastatic RCC treated for the first time with pazopanib. The study is designed to enroll approximately 700-1000 patients in over the course of an enrollment period of approximately 18 months. Sites will be contacted and qualified by the estimated number of advanced or metastatic RCC patients available for enrollment annually. To the extent possible, consecutive patients meeting inclusion/exclusion criteria will be enrolled. Sites will be required to maintain a patient enrolment log of eligible patients at their treatment centres. This log will document how patients came to be included or excluded from the study, in order to assess the representativeness of the study population. The overall number of patients and sites may be adjusted during the study to meet enrollment goals, if needed. Eligible patients will be enrolled by medical oncologists and potentially by urologists experienced in the management of patients with RCC, if consistent with local practice. There are no protocol-mandated visits or procedures associated with the study. Each patient is expected to participate for a maximum of 30 months or until premature discontinuation (i.e., due to death, withdrawal of consent, lost to follow-up or study termination). Follow-up information will be collected approximately every 3 months (a window of ± 4 weeks around the date of the suggested data collection will be allowed). If the patient is not seen for a regularly scheduled visit at that time, the site may contact the patient by telephone to solicit information regarding the events of interest and to limit loss to follow up. It is anticipated that frequency of patient assessment and imaging will differ according to local standard practice; therefore the quarterly data collection time points are intended to collect all assessments (with the date of assessment) since the previous visit date.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for enrolment in the study must meet all of the following criteria:

  * Age ≥ 18 years at enrollment
  * Documented diagnosis of advanced and/or metastatic clear cell or predominantly clear cell RCC
  * Clinical decision made to initiate treatment with pazopanib prior to enrollment in the study, but within 30 days of enrollment
  * Willing and able to provide written informed consent

Exclusion Criteria:

* Patients meeting any of the following criteria must not be enrolled in the study:

  * Patients currently participating in any interventional clinical trials in which treatment regimen and/or monitoring is dictated by a protocol
  * Previous exposure to an investigational or licensed multi-kinase inhibitor or an anti- VEGF angiogenesis inhibitor for advanced or metastatic disease
  * Life expectancy < 12 weeks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational studies plans to recruit from cliinics that are prescribing pazopanib to patients as part local standard of practice.
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2012-07-19 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | Approximately 30 months
  To evaluate overall survival (OS), progression-free survival (PFS) and the overall response rate (ORR) in patients treated with pazopanib
Relative Dose Intensity(RDI) | Approximately 30 months
  To characterize the relative dose intensity (RDI) and its observed effect on treatment outcomes
Characterise the RCC patient population treated | Approximately 30 months
  To characterise the RCC patient population treated with pazopanib (e.g., by demographics, disease characteristics, previous RCC treatment history) in comparison to a selected clinical trial population
Evaluate the change in health-related quality of life (HRQoL) | Approximately 30 months from baseline
  To evaluate the change in health-related quality of life (HRQoL) relative to baseline in patients treated with pazopanib
Evaluate Safety | From first treatment with pazopanib till 30 days after last dose of pazopanib treatment
  To evaluate the frequency of serious adverse events(SAEs) and adverse events of special interest (AESIs) in patients treated with pazopanib. Endpoint: Any adverse event that results in a pazopanib dose modification or discontinuation. Evidence of liver toxicity (e.g., increased ALT and/or AST, liver failure). New onset or worsened hypertension. Cardiac dysfunction (e.g., decreased left ventricular function, congestive heart failure). Thyroid dysfunction.

SECONDARY OUTCOMES:
Evaluate efficacy and safety comparable to VEG105192 | Approximately 30 months
  To evaluate clinical effectiveness, safety and RDI in those patients with comparable baseline characteristics to those included in the Phase III clinical trial [VEG105192]. Endpoints: Same as primary effectiveness, safety and RDI objectives
Evaluate efficacy, safety, RDI, and HRQoL | Approximately 30 months
  To evaluate clinical effectiveness, safety, RDI and HRQoL in relevant subgroups treated with pazopanib

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (126):
- United States (15):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Sioux Falls, South Dakota
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Houston, Texas
- Argentina (6):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, San Miguel de Tucumán
  - Novartis Investigative Site, Santa Fe
- Austria (8):
  - Novartis Investigative Site, Hall in Tirol
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, St.Veit/Glan
  - Novartis Investigative Site, Vienna
  - Novartis Investigative Site, Vöcklabruck
- Belgium (12):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Arlon
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Bouge
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Haine-Saint-Paul
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Ostend
  - Novartis Investigative Site, Ottignies
  - Novartis Investigative Site, Sint-Niklaas
  - Novartis Investigative Site, Verviers
- Colombia (3):
  - Novartis Investigative Site, Bucaramanga
  - Novartis Investigative Site, Medellín
  - Novartis Investigative Site, Montería
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Helsinki, Finland
- Germany (17):
  - Novartis Investigative Site, Kirchheim, Baden-Wurttemberg
  - Novartis Investigative Site, Aschaffenburg, Bavaria
  - Novartis Investigative Site, Erlangen, Bavaria
  - Novartis Investigative Site, Hof, Bavaria
  - Novartis Investigative Site, Landshut, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Lehrte, Lower Saxony
  - Novartis Investigative Site, Neubrandenburg, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Rostock, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Münster, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Homburg, Saarland
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Markkleeberg, Saxony
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Kiel, Schleswig-Holstein
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Hungary (6):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szombathely
  - Novartis Investigative Site, Veszprém
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Tel Aviv
- Italy (6):
  - Novartis Investigative Site, Napoli, Campania
  - Novartis Investigative Site, Modena, Emilia-Romagna
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Cremona, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Pavia, Lombardy
- Novartis Investigative Site, El Achrafiyé, Lebanon
- Novartis Investigative Site, Karachi, Pakistan
- Spain (25):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Albacete
  - Novartis Investigative Site, Badajoz
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Castellon
  - Novartis Investigative Site, Don Benito/Badajoz
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Guadalajara
  - Novartis Investigative Site, La Laguna (Santa Cruz de Tenerife)
  - Novartis Investigative Site, León
  - Novartis Investigative Site, Lleida
  - Novartis Investigative Site, Lugo
  - Novartis Investigative Site, Manresa (Barcelona)
  - Novartis Investigative Site, Ourense
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Sabadell (Barcelona)
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Santa Cruz de Tenerife
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Soria
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Valladolid
  - Novartis Investigative Site, Vigo ( Pontevedra)
  - Novartis Investigative Site, Zaragoza
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan Hsien
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kayseri
  - Novartis Investigative Site, Malatya
  - Novartis Investigative Site, Samsun
- United Kingdom (5):
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Shrewsbury

REFERENCES:
- [Derived] Procopio G, Bamias A, Schmidinger M, Hawkins R, Sanchez AR, Estevez SV, Srihari N, Kalofonos H, Bono P, Pisal CB, Hirschberg Y, Dezzani L, Ahmad Q, Rodriguez CS, Jonasch E. Real-world Effectiveness and Safety of Pazopanib in Patients With Intermediate Prognostic Risk Advanced Renal Cell Carcinoma. Clin Genitourin Cancer. 2019 Jun;17(3):e526-e533. doi: 10.1016/j.clgc.2019.01.018. PMID 31196680